CLINICAL TRIAL: NCT00438542
Title: HMW-Adiponectin is Raised in Newborns
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Other Study IDs: HMWadpkcb
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2007-02-22 (Estimated); Status verified 2007-02

CONDITIONS: Pre-Eclampsia
Keywords: Adiponectin, cord blood, pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Cross sectional, hospital-based study dealing with adiponectin levels in newborns to mothers with pre-eclampsia. Venus cord blood samples were collected immediately after birth; 30 cases and 62 controls were enrolled into the study. The study was approved by the local ethics committee and all participants gave written consent.

ELIGIBILITY:
Inclusion Criteria:

* Pre-eclampsia

Max Age: 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2003-07; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Lars Morkrid, MD, PhD, Study Director — Institute of Clinical Chemistry, Medical Faculty, University of Oslo, Norway